CLINICAL TRIAL: NCT01558986
Title: A Randomized, Double Blinded Placebo-Controlled Trial on the Routine Use of Preoperative Antibiotic Prophylaxis in Modified Radical Mastectomy
Brief Title: Routine Preoperative Antibiotic Prophylaxis in Modified Radical Mastectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of the Philippines (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NIH 2007-07-10-02
Record Dates: First submitted 2012-03-15; First posted 2012-03-20 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Surgical Infection
Keywords: Antibiotic prophylaxis; surgical site infection; modified radical mastectomy; Prevention of surgical site infection (SSI) in patients undergoing MRM for breast cancer
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Active Comparator): Patients to receive intravenous cefazolin 1 gram within 30 minutes prior to skin incision
  Interventions: Procedure: Cefazolin
- Placebo Arm (Placebo Comparator): Patients to receive sterile water only within 30 minutes prior to skin incision
  Interventions: Procedure: Sterile water

INTERVENTIONS:
Procedure: Cefazolin — Patients received intravenous cefazolin 1 gram within 30 minutes prior to skin incision;
  Arms: Treatment Arm
Procedure: Sterile water — Patients received sterile water only within 30 minutes prior to skin incision
  Arms: Placebo Arm

SUMMARY:
This is a randomized, double blinded, placebo-controlled trial on the routine use of preoperative antibiotic prophylaxis in modified radical mastectomy to evaluate the efficacy of preoperative prophylactic antibiotics in the prevention of surgical site infection (SSI) in patients undergoing modified radical mastectomy (MRM) for breast care.

DETAILED DESCRIPTION:
A randomized, double blinded, placebo-controlled trial on the routine use of preoperative antibiotic prophylaxis in modified radical mastectomy to evaluate the efficacy of preoperative prophylactic antibiotics in the prevention of surgical site infection (SSI) in patients undergoing modified radical mastectomy (MRM) for breast care.

Women with breast cancer who will undergo elective MRM were recruited for the study. Excluded were patients with significant co-morbid factors, for simultaneous breast reconstruction or bilateral oophorectomy, with intake of antibiotics within one week, with known allergy to cephalosporins, and those with local infection. Patients were randomized to receive either transvenous cefazolin 1 gram or sterile water only within 30 minutes prior to skin incision. Standard skin preparation and operative technique for MRM were carried out. Wounds were assessed for the presence of SSI and other complications weekly for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically diagnosed breast cancer of age group 18-80 years old, ECOG 0-1, clinical stage I to IIIB, admitted to the surgery ward, who were scheduled for elective MRM.

Exclusion Criteria:

* Women with significant co-morbid factors (diabetes mellitus, severe malnutrition, corticosteroid therapy), those scheduled for simultaneous breast reconstruction or bilateral oophorectomy, with intake of antibiotics within one week prior to surgery, with known allergy to cephalosporins, and those with local infection.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2007-12; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Surgical Site Infection (as defined by the Centers for Disease Control and Prevention) | Wounds were assessed on the first post-operative day, then patients were followed-up every week after discharge for the duration of 30 days
  Mastectomy wounds were evaluated for the presence of SSI as defined by the Center for Disease Control and Prevention meeting the following criteria: infection that occurred within 30 days after the operative procedure and at least one of the following:
  1. purulent drainage (culture documentation not required)
  2. organism isolated from fluid/tissue of incision site
  3. at least one sign of inflammation (erythema, local warmth of wound, induration)
  4. wound is deliberately opened by the surgeon
  5. physician declares the wound infected

CONTACTS AND LOCATIONS:
Overall Officials: Nelson C Cabaluna, Doctor of Medicine, Principal Investigator — University of the Philippines Manila
Locations (1):
- Philippine General Hospital - University of the Philippines Manila, Manila, Philippines

REFERENCES:
- [Derived] Cabaluna ND, Uy GB, Galicia RM, Cortez SC, Yray MD, Buckley BS. A randomized, double-blinded placebo-controlled clinical trial of the routine use of preoperative antibiotic prophylaxis in modified radical mastectomy. World J Surg. 2013 Jan;37(1):59-66. doi: 10.1007/s00268-012-1816-5. PMID 23052809